CLINICAL TRIAL: NCT05917535
Title: Mentalizing Education in a Psychiatric Out-patient Clinic in North Norway
Brief Title: Mentalizing Education in a Psychiatric Out-patient Clinic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Principal Investigator, Poul Lundgaard Bak, Principal Investigator, University Hospital of North Norway
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: DPSHA-UNN Mz Study
Record Dates: First submitted 2023-03-14; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-03

CONDITIONS: Mental Health Education

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients offered mentalizing course supplemental to treatment as usual
  Interventions: Behavioral: Mentalizing course
- Control (No Intervention): Control group - treatment as usual.

INTERVENTIONS:
Behavioral: Mentalizing course — 6 hour mental health education course about mentalizing.
  Arms: Intervention group

SUMMARY:
Mentalization-based Mental Health Education in a naturalistic patient population from a psychiatric out-patient clinic in North Norway: A randomized controlled study

DETAILED DESCRIPTION:
Half of an unselecected waiting list group of patients (randomized) from a psychiatric out-patient clinic are offered a 6 hour mental health education course abour mentalizing. 1 year follow up period. Primary outcome variable is use of hospital services. Secondary outcome variables are questionnaire scores.

ELIGIBILITY:
Inclusion Criteria:

* all norwegian speaking patients referred to the outpatient clinic

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Hospital service us | 1year
  Contact days (policlinic, inpatient ward and emergency team)

SECONDARY OUTCOMES:
3 item wellbeing questionnaire | 6 month
  Each question is answered on a separate 0-9 point scale. Higher scores means better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Poul Lundgaard, MD, Principal Investigator — University Hospital North Norway
Locations (1):
- University Hospital North Norway, Harstad, Norway

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/35/NCT05917535/Prot_000.pdf